CLINICAL TRIAL: NCT02219776
Title: Decreasing Proprionbacterium Acne Skin Colonization Prior to Arthroscopic Shoulder Surgery
Brief Title: Decreasing Infection In Arthroscopic Shoulder Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McLaren Health Care (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 201400113
Record Dates: First submitted 2014-08-16; First posted 2014-08-19 (Estimated); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Post Operative Infection Arthroscopic Shoulder Surgery; Infection
Keywords: Infection,; Proprionbacterium Acne,; Shoulder,; skin preparation
MeSH Terms: conditions — Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chlorhexidine Standard of Care Arm (Active Comparator): Use of Chlorhexidine to cleanse pre-operative surgery site
  Interventions: Other: Standard of Care - Chlorhexidine Scrub only
- Benzoyl Peroxide Experimental Arm (Experimental): Use of Chlorhexidine scrub brush and 1.5 oz bottle of 10% benzoyl peroxide emollient
  Interventions: Drug: Benzoyl Peroxide solution Plus Chlorhexidine Scrub

INTERVENTIONS:
Drug: Benzoyl Peroxide solution Plus Chlorhexidine Scrub — Subjects will be provided instructions on how to use and apply the chlorhexidine using a scrub brush and 1.5 oz bottle of 10% benzoyl peroxide emollient application
  Arms: Benzoyl Peroxide Experimental Arm
Other: Standard of Care - Chlorhexidine Scrub only — Subjects will be given instructions on how to apply the Chlorhexidine using a scrub brush
  Arms: Chlorhexidine Standard of Care Arm

SUMMARY:
Despite the use of a standard preoperative skin disinfectant prior to shoulder surgery propionibacterium acne remains a leading cause of post-operative infections. The purpose of this study is to evaluate effectiveness of topical benzoyl peroxide as an adjuvant to chlorhexidine-impregnated skin preparation in attempting to lower the colonization propionibacterium acne prior to surgery. This study will take cultures from patients who are randomly assigned into groups that receive and do not receive benzoyl peroxide as additional skin prep prior to elective shoulder surgery and compare quantified culture results.

DETAILED DESCRIPTION:
With IRB approval and informed consent to participate in the study, patients scheduled for elective shoulder arthroscopy will be randomly selected and placed into 1 of 2 groups. Both groups will adhere to the surgeon's preoperative protocol of showering the night before with instructions to scrub the operative shoulder including the axilla with a chlorhexidine scrub brush. Group 1 will be treated "per protocol" and only be given instructions to use chlorhexidine. While group 2 will be provided a chlorhexidine scrub brush and a 1.5oz bottle of 10% benzoyl peroxide emollient to be applied after using the chlorhexidine scrub. The benzoyl peroxide should not be washed off prior to surgery.

Thirty minutes prior to incision, intravenous antibiotics, cefazolin or clindamycin if penicillin intolerant, will be administered per protocol. Dry anaerobic culturettes will be taken at the location of the expected posterior portal location before and after the application of the chloraprep solution. At the time of surgery both groups will undergo preoperative skin preparation, in sterile fashion, with our institutions "standard" protocol utilizing ChloraPrep (2% chlorhexidine gluconate and 70% isopropyl alcohol; Enturia, El Paso, Texas). In addition, a 3mm full thickness skin punch biopsy will be taken after, application of chlorprep. Biopsies will be immediately placed, by the surgeon, in sterile receptacle with sterile saline and sent to our microbiology department. The biopsy site will be incorporated into the portal incision and will be closed appropriately minimizing the morbidity of obtaining the biopsy.

The culture results will be recorded into a "dummy" account on McLaren's electronic medical records program. This account ensures that the costs of the study are not charged to the patient as well as blinding the patient and surgeon of the their results. The patient correlating information will only be known to Dr. Fine and they will be kept in a password protect computer document which will be kept in a off campus protected locked location.

The Microbiology lab will place the swab specimens in 1 ml of saline, vortex them, and inoculate 0.01 mL onto an anaerobic blood agar plate. A chopped meat broth will also be inoculated. The punch biopsies will be ground and then inoculated to an anaerobic blood agar plate and a chopped meat broth. The anaerobic plates will be incubated in an anaerobic chamber at 35°C. The plates and broth will be examined daily for the first 4 days, then on days 7, 10 and 14 and any growth screened to determine if P. acnes is present. Results will be reported as "no P. acnes isolated" or as "<X>CFU/mL P. acnes" for the swab specimens. No colony count can be issued for the biopsies. These will be reported semi-quantitatively as rare, few, moderate or many. All plates will be read and counted manually by a laboratory technician who is not involved in the study and has been blinded from preoperative prep used. If any growth is detected, the sample will be considered positive.

ELIGIBILITY:
Inclusion criteria:

1. Elective arthroscopic shoulder surgery
2. Ages > 18
3. Male and Female

Exclusion criteria:

1. Active Infection
2. History of ipsilateral prior shoulder surgery
3. History of prior shoulder infection
4. Current use of Antibiotics
5. History of immunosuppression
6. Open wounds
7. History of Inflammatory arthritis
8. Allergy to benzoyl peroxide
9. Allergy to chlorhexidine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-09; Primary Completion 2021-06 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
Bacterial Growth | 14 days from culture
  Skin swabs and biopsy will be cultured for 14 days in media specific for growing P.Acne

CONTACTS AND LOCATIONS:
Overall Officials: Landon R Fine, DO, Principal Investigator — McLaren Greater Lansing
Locations (1):
- McLaren Greater Lansing, Lansing, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided